CLINICAL TRIAL: NCT06055634
Title: SIRT1(rs7069102 ) Gene Polymorphism in Chronic Obstructive Pulmonary Disease at Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Kadry, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-09-10PD
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Genotyping of SIRT1in Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients more than 40 years
  Interventions: Genetic: genotyping of SIRT1 in chronic obstructive patients
- patients less than 40 years
  Interventions: Genetic: genotyping of SIRT1 in chronic obstructive patients
- controls
  Interventions: Genetic: genotyping of SIRT1 in chronic obstructive patients

INTERVENTIONS:
Genetic: genotyping of SIRT1 in chronic obstructive patients — genotyping of SIRT1 in chronic obstructive patients

SUMMARY:
Chronic obstructive pulmonary disease (COPD) prevalence, morbidity, and mortality vary across countries and across different groups within countries with a direct relation to the prevalence of tobacco smoking. Other risk factors for COPD include genetic factors, longstanding asthma, outdoor air pollution, second-hand smoke exposure, biomass smoke, indoor air pollution, occupational exposures, and tuberculosis . The prevalence and burden of COPD are projected to increase in the coming decades because of continued exposure to COPD risk factors and the changing age structure of the world's population. As these factors are rapidly increasing in developing countries, COPD will become a major health problem, exerting a huge demand on economic and healthcare resources in developing countries [2]. In Egypt, although COPD is a rising significant health problem, data on its prevalence, morbidity, and mortality are still lacking and have to be estimated .

Sirtuin 1 (SIRT1) is a protein/histone deacetylase dependent NAD. It plays a crucial role in various human diseases such as cardiovascular diseases, cancer, inflammation, aging, neurodegenerative disease, obesity and type 2 diabetes. Seven isoforms of the SIRT1 gene (SIRT1- SIRT7) have been determined in mammals. Expression of the SIRT1 gene is regulated by transcription factors such as CREB, FOXO3, HIC1, NF-KB, p53, PARP-2 and PPAR. SIRT1

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Sohag University Hospital, chest department.

Exclusion Criteria:

* Patients with malignancies, any other chronic disease, Individuals with a history of known chronic cardiorespiratory diseases and those with collagen vascular diseases were excluded.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 100 individuals at high risk for COPD were studied from approval of the ethical committee of the Faculty of Medicine, Sohag University. Informed consent was obtained from all participants. 100 healthy control.
  All participants will subject to the following: (1) A questionnaire including age, sex, smoking status, presence of chronic cough, chronic sputum production, chest wheezing, and shortness of breath; grading of dyspnea using a modified medical research council (MMRC) dyspnea scale. (2) General examination, including measurements of body weight, height, and BMI. (3) Local chest examination.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
SIRT1(rs7069102 ) Gene polymorphism in chronic obstructive pulmonary disease | 2 months
  genotyping of sirt1 in chronic obstructive pulmonary disease

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eisner MD, Anthonisen N, Coultas D, Kuenzli N, Perez-Padilla R, Postma D, Romieu I, Silverman EK, Balmes JR; Committee on Nonsmoking COPD, Environmental and Occupational Health Assembly. An official American Thoracic Society public policy statement: Novel risk factors and the global burden of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 Sep 1;182(5):693-718. doi: 10.1164/rccm.200811-1757ST. PMID 20802169
- [Background] Chan-Yeung M, Ait-Khaled N, White N, Ip MS, Tan WC. The burden and impact of COPD in Asia and Africa. Int J Tuberc Lung Dis. 2004 Jan;8(1):2-14. PMID 14974740
- [Background] Zarrabeitia MT, Valero C, Martin-Escudero JC, Olmos JM, Bolado-Carrancio A, de Sande-Nacarino EL, Rodriguez-Rey JC, Sainz J, Riancho JA. Association study of sirtuin 1 polymorphisms with bone mineral density and body mass index. Arch Med Res. 2012 Jul;43(5):363-8. doi: 10.1016/j.arcmed.2012.06.012. Epub 2012 Jul 21. PMID 22824213
- [Background] Rahman I, Kinnula VL, Gorbunova V, Yao H. SIRT1 as a therapeutic target in inflammaging of the pulmonary disease. Prev Med. 2012 May;54 Suppl(Suppl):S20-8. doi: 10.1016/j.ypmed.2011.11.014. Epub 2011 Dec 8. PMID 22178470